CLINICAL TRIAL: NCT03544788
Title: HEAL I (The Treatment of Venous Leg Ulcers): Evaluation of Cirvo™ Mobile Compression Device for the Treatment of Venous Leg Ulcers
Brief Title: Evaluation of Cirvo™ Mobile Compression Device for Treatment of Venous Leg Ulcers
Acronym: HEAL I
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Business decision
Sponsor: Radial Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RMP-002
Record Dates: First submitted 2018-05-21; First posted 2018-06-04 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Venous Leg Ulcer
Keywords: mobile compression device
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Intervention Model Description: Cirvo™ Therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Cirvo™ Therapy (Experimental)
  Interventions: Device: Cirvo™ Therapy

INTERVENTIONS:
Device: Cirvo™ Therapy — The Cirvo(TM) (also referred to as the Radial Medical Compression System) is a mobile wearable medical device that applies graded intermittent mechanical sequential compression for the treatment of venous leg ulcers (VLU).

SUMMARY:
This study in venous leg ulcer (VLU) patients will evaluate the use of Cirvo™ therapy for the treatment of VLU when applied for a minimum of two hours daily for up to 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients between 18 and 80 years of age
2. Patients (CEAP 6) who have not previously experienced a period of open ulceration exceeding 26 weeks in the affected leg
3. Total venous ulcer area < 20cm2
4. Duration of therapy for active venous ulcer <26 weeks prior to enrollment
5. Venous insufficiency documented by venous reflex ultrasound showing mild, moderate, or severe reflux in the superficial or deep venous system

Exclusion Criteria:

1. Acute DVT within the 3 months prior to enrollment
2. Ulcer present for <2 weeks
3. Ulcers extending with exposed fascia, tendon, or bone within the wound margins
4. Lateral malleolus ulcers
5. Ulcers with perforator incompetence deep to the ulceration (within 5 cm of the wound border)
6. Active infection (systemic or in the affected limb)
7. Lower extremity gangrene
8. Diabetes mellitus (Type I or II) requiring medication
9. History of pulmonary vascular disease (PVD)
10. History of pulmonary edema
11. History of decompensated congestive heart failure (CHF)
12. Open surgery or major trauma to the legs within the last six months
13. History of lower limb malignancy, primary or secondary
14. Acute symptomatic lower extremity thrombophlebitis
15. Pregnant or breastfeeding
16. Calf geometry on which Cirvo(TM) device does not appropriately fit
17. Known sensitivity to any of the materials used in the Cirvo(TM) device
18. Currently participating or plans to participate in in any other investigational clinical evaluation during the 12 week study period that may, in the opinion of the investigator, affect blood flow and/or venous leg ulcer

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06-30 (Estimated); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
Percent of subjects fully healed at 12 weeks | 12 weeks

SECONDARY OUTCOMES:
Percent of wound epithelialized at 12 weeks | 12 weeks
Percent of subjects fully healed at 4 weeks | 4 weeks

OTHER OUTCOMES:
Time to complete healing in fully-healed subjects | 12 weeks
Therapy-related adverse events will be collected throughout the 12-week study period | 12 weeks
Characterization of Quality of Life measured using the EQ-5D-5L | Baseline, 4 weeks, 12 weeks
Characterization of Quality of Life measured using the WPAI:GH | Baseline, 4 weeks, 12 weeks
  WPAI:GH: Work Productivity and Activity Impairment: General Health
Characterization of Disability measured using the VLU-QoL | Baseline, 4 weeks, 12 weeks
  VLU-QoL: Venous Leg Ulcer Quality of Life Instrument
Characterization of Disability measured using the VCSS | Baseline, 4 weeks, 12 weeks
  VCSS: Venous Clinical Severity Score
Characterization of Patient Satisfaction measured using a Patient Satisfaction Survey | Baseline, 4 weeks, 12 weeks
Measurement of compliance with Cirvo(TM) (a minimum of 2 hours of therapy daily for up to 12 weeks) - number of days of therapy use | 12 weeks
Measurement of compliance with Cirvo(TM) (a minimum of 2 hours of therapy daily for up to 12 weeks) - hours per day of therapy use | 12 weeks
Reasons for Cirvo(TM) discontinuation prior to complete healing (including, but not limited to: adverse events, self-withdrawal) will be tabulated | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Zuckerberg San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No